CLINICAL TRIAL: NCT04021095
Title: An Exploratory Study on the Development of a Novel Head Protection Prototype Device for Post-decompression Craniectomy Patients
Brief Title: Novel Head Protection Prototype Device for Decompression Craniectomy
Acronym: HPPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: Creatz3D (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DSRB2019/00155
Record Dates: First submitted 2019-07-11; First posted 2019-07-16 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2019-11

CONDITIONS: Brain Injuries; Stroke
MeSH Terms: conditions — Brain Injuries; Stroke

STUDY DESIGN:
Intervention Model Description: Customised head protection prototype device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Decompressive craniectomy (Experimental): 3D printed skull replacement piece will be fitted to subject.
  Interventions: Device: Head protection prototype device

INTERVENTIONS:
Device: Head protection prototype device — The proposed experimental HPPD uses biocompatible material using FDMÔNylon which has high fatigue resistance, chemical resistance with impact resistance and toughness which is free of powders. It is HSA unclassified as yet and the FDMONylon is not FDA approved yet.

SUMMARY:
A proof-of-concept (POC) proposal to study the feasibility of customized head protection prototype device (HPPD) using 3D printed externally-applied moulded skin prosthesis integrated to the craniectomy bony skull defect.

DETAILED DESCRIPTION:
A proof-of-concept (POC) proposal to study the feasibility of customized head protection prototype device (HPPD) using 3D printed externally-applied moulded skin prosthesis integrated to the craniectomy bony skull defect. The proposed material is a bio-compatible, light-weight rigid /semi rigid material which can be fitted to the skull defect and interfaced with the subject's bony rim using soft, deformable material (e.g. silicon) and attached using an elastic head band or other acceptable means. The prosthesis is removable for skin and prosthesis cleansing and ventilation.

Study Specific Objectives:

(i) Primary Objectives

These are to:

1. test the feasibility and safety of customised 3D printed HPPD,
2. integrate the prostheses to the skull defect in removable manner and discharge patient with appropriate education,
3. to systematically monitor subjects for symptoms, compliance, complications and subjective feedback during the outpatient phase where progressive wear of HPPD and monitoring of acceptability will be monitored.

ELIGIBILITY:
Inclusion Criteria:

All subjects must meet all of the inclusion criteria to participate in this study.

1. Age 21 to 80 years, both males and females.
2. Presence of surgical unilateral or bilateral craniectomy performed for reasons of ischaemic or haemorrhagic stroke, Subarachnoid haemorrhage (SAH), traumatic brain injury (TBI), benign cerebral tumours, etc.
3. Stroke, SAH or TBI are diagnosed by specialists and confirmed on brain imaging studies (CT, MRI)
4. Duration from event > 30 days and either during inpatient or outpatient phase.
5. Presence of at least 1 post decompressive craniectomy CT brain film performed at NNI/TTSH.
6. Healed craniectomy surgical wound without bulging skin flap or active skin infection.
7. Patients awaiting elective cranioplasty or those who refuse cranioplasty. 8 Ability to understand simple instructions and give own consent. 9 Presence of family members or NOK who can supervise the patient to don the head protection device, care for the material and regularly monitor for compliance and complications 10 Reproductive age females should not be pregnant at the point of consent-taking and during the study

Exclusion Criteria:

1. Patient in vegetative or minimally responsive state.
2. Presence of uncontrolled medical condition (uncontrolled hypertension, Diabetes Mellitus, sepsis or delirium, active malignancy either cranial or extracranial sites)
3. Presence of end organ failure (end stage renal or liver failure, renal dialysis, life expectancy <6 months)
4. Presence of pregnancy or lactation.
5. Presence of severe agitation /behavioural/active depression or anxiety/ drug or alcohol addiction which would negatively affect compliance,
6. Presence of unhealed head wound, active wound infection, scalp dermatitis, wound breakdown which would be worsened by pressure from the HPPD.
7. Presence of known allergy to the investigational products which is the 3D printed material (e.g. Nylon).
8. Subjects' CT brain imaging films are not available to the study team.
9. Absence of NOK who can assist monitoring unless subjects is able to self-monitor

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-07-04 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Percentage of acute complications at second hour of HPPD fitting | 12 months
  Complications are defined as immediate complaints of pain or discomfort and /or signs of bony defect scar pressure redness or wound breakdown within the first 2 hours in the research clinic.

SECONDARY OUTCOMES:
Percentage of acute complications at end of first week of HPPD use. | 12 months
  Complications are defined as pain or discomfort or signs of bony defect scar pressure or redness or wound breakdown in the first week post-fitting of HPPD

CONTACTS AND LOCATIONS:
Overall Officials: Khai Pang Leong, Study Director — Tan Tock Seng Hospital Clinical research and innovation office
Locations (1):
- Tan Tock Seng Hospital Rehabilitation Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Due to the visual nature of the study data (digital photo facial images), only study team researchers will have access to identifiable participant data and images.